CLINICAL TRIAL: NCT06667791
Title: Evaluation of Computer-guided Visco Supplementation in the Management of Internal Derangement of Temporomandibular Joint (a Randomized Controlled Clinical Trial)
Brief Title: Computer Guided Visco Supplementation in the Management of Internal Derangement of Temporomandibular Joint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant Lecturer of Dental Public Health and biostatistical consultant, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0870-04
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Temporomandibular Disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental)
  Interventions: Other: Computer guided sodium hyaluronate injections
- Control (Active Comparator)
  Interventions: Other: conventional sodiumhyaluronate injections

INTERVENTIONS:
Other: Computer guided sodium hyaluronate injections — Patients will be treated with Computer guided sodium hyaluronate injections in superior TMJ space
  Arms: Study Group
Other: conventional sodiumhyaluronate injections — Patients will be treated with conventional sodium hyaluronate injections in superior TMJ space
  Arms: Control

SUMMARY:
Background: The intra-articular injection is considered the first line of minimally invasive treatment in TMJ-ID patients who do not respond to conservative treatment. Image-guided puncture technique has emerged to add safety, reliability, convenience, and decrease the need for correcting the puncture point.

Aim of the study: To evaluate the feasibility and clinical outcomes of computer-guided superior joint space injection of sodium hyaluronate in the treatment of temporomandibular joint disorder (TMJ-ID) compared with conventional injection

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients diagnosed with internal derangement according to Wilkins stage I and II.
* Patients who would not respond to conservative treatment as a first line of treatment.

Exclusion Criteria:

* Patients with Wilkins stage III, IV, V.
* History of mandibular fracture.
* Lactating, pregnant or planning pregnancy women.
* Known hypersensitivity to hyaluronic acid or clear biocompatible photopolymer resin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-05-03 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
Change in TMJ dysfunction | Baseline, 1 month, and 3 months
  A modified version of Helkimo's clinical dysfunction index (Di) is be calculated to assess the TMJ dysfunction as follows:
  * Maximum unassisted mouth opening range: Opening range will be determined by asking the patient to gently open mouth and measure the distance between upper and lower central incisors.
  * Mandibular deviation during opening: Patients will be asked to open mouth gently and deviation will be noted between maxillary and mandibular midline, score 0 - if <2 mm, score 1 - if 2-5 mm, and score 5 - if >5 mm
change in pain score | Baseline,1 months, and 3 months
  Pain level was determined by the patient's self-assessment using a visual analog scale (VAS) from zero to 10 ("0" is pain-free and "10" is severe intolerable pain).

SECONDARY OUTCOMES:
Duration of operation | Baseline
  Total procedural time consumed starting from the application of topical antiseptic up to the end of the procedure.
Number of Needle Relocation | Baseline
  The need to relocate the needle after first puncture of both needles will be used to compare between the efficacies of the computer guided arthrocentesis guide and the conventional free hand arthrocentesis.

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient clinic of Oral and Maxillofacial Surgery, Alexandria, Egypt